CLINICAL TRIAL: NCT05631522
Title: The Effect of Foot Reflexology on Pain Severity Associated With Mediastinal Chest Drain Removal in Patients Undergoing Open-Heart Surgery
Brief Title: Effect of Foot Reflexology on Pain Associated With Mediastinal Chest Drain Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, afnan attia ibrahim mohamed, demonstrator of critical care and emergency nursing, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P.0235
Record Dates: First submitted 2022-05-26; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Foot Reflexology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot reflexology group (Experimental): Patients who will receive foot reflexology before and throughout the MCDR procedure.
  Interventions: Other: foot reflexology
- control group (No Intervention): Patients who will receive the routine ICU care during the MCDR procedure.

INTERVENTIONS:
Other: foot reflexology — Warm-Up Phase:
  Pre-reflexology foot massage and all-over foot squeeze will be performed for two minutes.
  Mini-Reflexology Session:
  Specific reflexology will be performed with special attention to two important foot reflex areas that include:
  Diaphragm and Solar Plexus Reflex Areas are located in the distance between the upper and middle third of the sole.
  The Heart and Lung Reflex Areas are located below the chest of the foot. The heart pumps the oxygen-rich blood around the body
  Arms: foot reflexology group

SUMMARY:
Cardiovascular diseases (CVDs) remain the leading cause of death worldwide and significantly affect patient quality of life and socioeconomic status. The care of CVD patients in Egypt is very complex and sensitive because of the high incidence and high mortality rate. The burden of CVD and the high prevalence of CVD risk factors in Egypt are alarming.

Despite great evidence of adverse clinical impact, the pain remains infrequently assessed and poorly managed in ICU. Pain has serious physical and psychological effects which can impair patient recovery and discharge. Moreover, it does not allow the patients to collaborate appropriately during care-related procedures, such as mobilization and respiratory therapy.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a general term for conditions affecting the heart or blood vessels. It is commonly associated with an increased risk of blood clots and build-up of fatty deposits inside the arteries. CVD is the leading global cause of death accounting for more than 17.9 million deaths per year in 2019, representing 32% of all global deaths. Of these deaths, 85% were due to heart attack and stroke (World Health Organization [WHO], 2021). Mortality rate due to CVD is expected to grow to more than 23.6 million by 2030 (American Heart Association [AHA], 2017). In Egypt, the CVD mortality rate accounts for 46% of total deaths from all ages for both sexes (WHO, 2014).

There are many options for treating CVD, one of these options is open-heart surgery (OHS) especially coronary artery bypass graft (CABG) and valvular surgeries. CABG is done in patients with severe narrowing of the coronary arteries that do not respond to other treatment. Patients after OHS are usually transferred to the intensive care unit (ICU) to receive advanced medical care and close monitoring. They may suffer pain after OHS for various reasons including sternum incision, tissue excision, removal of saphenous vein, and the presence of chest drain as well as various factors related to the type of operation). Patients in the ICU are also exposed to many invasive and noninvasive painful procedures for diagnostic or therapeutic purposes.

Mediastinal chest drain placement (MCDP) and removal is one of these painful procedures. MCDP is a part from the standard care in cardiac surgery to assist the clearance of blood from the pericardial space. The mediastinum is the region between the pleural sacs, containing the heart and all of the thoracic viscera except the lungs. Drainage of fluid, or blood from the pericardial space after OHS is necessary to prevent complications as pericardium effusions and cardiac tamponade. It also helps to detect hemorrhage. Therefore, negative pressure drain is placed in the mediastinum .

Cardiac tamponade may occur after OHS as a result of blood or fluid collecting in the pericardial space compressing the heart and reducing cardiac output. However, mediastinal chest drain removal (MCDR) is a standardized potentially painful procedure that is commonly associated with pain and can be the worst hospital experience for those patients. MCDP after OHS is traditionally achieved using large-bore (28-36 Fr) plastic chest tubes for the first 24 hours after surgery or until drainage is minimal. MCDR reduces pain and improves the forced expiratory volume in one second. Therefore, it can improve the patients' fast recovery.

Separation of the drain from the adjoined tissues is painful as it adheres to the surrounding tissues. Sternal pain is a prevalent complication caused by CABG, which normally initiates within a few hours after surgery, and with poor control it is likely to predispose the patients to chronic pains lasting for six months to one year postoperatively.

The most disturbing complaint after OHS is acute pain, which is still a severe and under-treated problem. Moreover, MCDR is described as the worst pain experienced during the first 48 hours, which are spent in the ICU. Sternal pain may occur due to changing positions, coughing, deep breathing, use of a spirometer and movement in bed.

As being the fifth vital sign, pain is one of the most important factors causing physical and psychological discomfort to patients in the ICU. It induces physiological changes in most organ systems (WHO, 2011). Pain is a common symptom that increases patients' suffering and prolongs their hospital stay. This can delay their recovery time as the physiologic responses to pain inhibit the body's ability to react positively during the healing process.

Pain in ICU patients can contribute to unfavorable outcomes. The stress response to pain may cause hyperglycemia and increase catecholamine, cortisol, and antidiuretic hormone secretions. In addition, pain-induced reflex responses may alter respiratory mechanics, increase cardiac demands, and cause muscle spasms, rigidity, and contraction of skeletal muscles. There are many available pain assessment tools. These tools are used according to the patient's condition. If the patient is conscious and able to self-report pain, a visual analog scale and numerical rating scale can be used . For unconscious patients; a behavioral pain scale or the critical care observation tool can be used.

Pain management aims to alleviate pain or reduce it to an acceptable level. It includes two main basic approaches: pharmacological and non-pharmacological measures. Pharmacologic pain management refers to the use of medications as narcotics and non-narcotics analgesics. These medications control pain effectively but may be associated with many physical and psychological side effects. Additionally, the risk of drug dependency is high and the drugs are expensive. Moreover, using analgesics is the most common method to alleviate the pain induced by MCDR, but the patient response to medication can vary and may not achieve complete relaxation.

While non-pharmacological pain management measures include local anesthesia and complementary therapy. A combination of pharmacological and non-pharmacological approaches is reported to achieve the highest level of pain control with the least complications. Complementary therapy includes relaxation, touch therapy, music therapy, imagination, self-management, social support, and applying hot and cold therapy.

New modalities such as reflexology and cryotherapy can be used to deal with patients' pain, stress, and anxiety. These methods are simple, less expensive, non-invasive, and with fewer side effects. Reflexology is one of the most common complementary therapy used to produce stimulations on the referred reflexology areas. It is a systematic technique of applying pressure to particular points on the feet and hands to impact the health of related parts of the body. Each pressure point acts as a sensor that is linked with specific parts of the body. There are reflex points or zones in the feet correlated with all body parts. These zones form a chart of the body in the feet. Hence, when a specific reflex area is excited, the cells of the body comply by creating a reflex effect on the corresponding organs, nerves, tissues, and muscles.

Foot reflexology has been found to have the greatest impact on patients after cardiac surgery. It reduces tension, relieves fatigue, improves sleep and recovery time. It also reduces pain levels in patients following cardiac surgery. Evidence shows that reflexology massage is a simple and cost-effective technique. Moreover, it is considered a non-invasive method used to regulate the activity of the autonomic nervous system, coordinate physiological responses, alleviate anxiety, and induce relaxation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult conscious patients ≥ 18 years old after OHS, who have a mediastinal chest drain.
2. Gender: male and female

Exclusion Criteria:

- 1. Sedated patients 2. Patients with any problem in the foot as a wound, allergy, injury, pain, callus, corn, fungal skin infection, or previous scars.

3. Patients use analgesics for 6 hours before the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Efficacy of foot reflexology on pain | 1 day
  Incidence of pain during chest drain removal. Pain assessed by NRS [The scoring system is interpreted as 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain] and CPOT scale [This pain assessment tool evaluates four clinical components: facial expressions, body movements, muscle tension, and compliance with the ventilator for mechanically ventilated patients or vocalization for the non-intubated patients. The CPOT score ranges from 2 to 8 and a score of more than 2 require pain management].